CLINICAL TRIAL: NCT02811406
Title: The Role of Intravenous Albumin Replacement During Abdominal Paracentesis in Patients With Malignancy Related Ascites
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MC01/02/16; 2016/00326 (Other: NHG DSRB)
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Ascites; Hypotension
MeSH Terms: conditions — Ascites; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receives IV albumin infusion (Experimental): IV albumin 20% 50 mL for every 1L of ascitic fluid drained
  Interventions: Procedure: Receives IV albumin infusion
- Do not receive IV albumin infusion (Placebo Comparator): No IV albumin infusion
  Interventions: Biological: Do not receive IV albumin infusion

INTERVENTIONS:
Procedure: Receives IV albumin infusion — IV albumin 20% 50 mL for every 1L of ascitic fluid drained. Blood pressure and heart rate are recorded every four hours in both groups in the first 48 hours.
  If hypotension occurs (defined as fall in systolic blood pressure of > 20 mmHg from baseline) during drainage, drain is clamped and the patient will be clinically evaluated for cause of hypotension. If no other causes of hypotension are found and patient remains asymptomatic, repeat blood pressure measurement in 30 minutes. If blood pressure maintains > 90/50 mmHg after 30 minutes and patient is asymptomatic, continue drainage and patient stays in the study. If patient remains hypotensive (BP < 90/50) or develops symptomatic hypotension, then the patient will be taken off study and the hypotension managed as clinically indicated.
  Arms: Receives IV albumin infusion
Biological: Do not receive IV albumin infusion — No IV albumin infusion. Blood pressure and heart rate are recorded every four hours in both groups in the first 48 hours.
  If hypotension occurs (defined as fall in systolic blood pressure of > 20 mmHg from baseline) during drainage, drain is clamped and the patient will be clinically evaluated for cause of hypotension. If no other causes of hypotension are found and patient remains asymptomatic, repeat blood pressure measurement in 30 minutes. If blood pressure maintains > 90/50 mmHg after 30 minutes and patient is asymptomatic, continue drainage and patient stays in the study. If patient remains hypotensive (BP < 90/50) or develops symptomatic hypotension, then the patient will be taken off study and the hypotension managed as clinically indicated.
  Arms: Do not receive IV albumin infusion

SUMMARY:
Aims: To compare the rates of hypotension in patients with malignancy-related ascites undergoing abdominal paracentesis with and without prophylactic intravenous albumin infusion

Methodology: Patients with symptomatic ascites secondary to underlying malignancy admitted to medical oncology inpatient service who require abdominal paracentesis will be enrolled. Patients with known portal hypertension based on SAAG (>11.1 mmol/L) will be excluded. Eligible patients are randomized 1:1 to two groups. During drainage of ascites fluid, one group will receive intravenous albumin infusion (50 ml/Litre of ascitic fluid drained), whereas the other group will not receive intravenous albumin infusion. Baseline parameters along with routine 4 hourly monitoring of blood pressure will be done. Episodes of hypotension (fall in SBP > 20 mmHg) will be compared between these two groups and significance tested using the chi-square test.

Clinical significance: Ascites often occurs in the setting of advanced malignancy and drainage of ascites has been proven to provide symptomatic relief in this patient population with relatively short life expectancy. The use of intravenous albumin infusion is loosely extrapolated from studies in patients with liver cirrhosis undergoing abdominal paracentesis. To date, there have been no standard guidelines to guide practice and no studies looking at the use of intravenous albumin in this population. As the mechanisms of ascites are different in different malignancies, the indication of intravenous albumin is uncertain and perhaps unnecessary in this setting. We hope to understand more about the rates of hypotension during abdominal paracentesis in this population and to generate systematic data to guide clinical practice in this area.

DETAILED DESCRIPTION:
General Introduction:

Therapeutic paracentesis is the first line of treatment for patients with symptomatic malignant ascites. The practice of intravenous albumin infusion during abdominal paracentesis comes from evidence in patients with liver cirrhosis. A meta-analysis of seventeen randomised trials evaluating patients receiving albumin versus alternative treatment during large volume paracentesis found that albumin reduced the incidence of post-paracentesis circulatory dysfunction, hyponatraemia and mortality (Bernardi M, 2012). The mechanisms of ascites in patients with cirrhosis are driven by portal hypertension. Portal hypertension brings about systemic vasodilation and hyperdynamic circulation that eventually contribute to functional and biochemical changes leading to ascites (Gines. P, 1997).

In contrast, cause of ascites in patients with malignancies is usually multi-factorial. It occurs commonly in several tumours including malignancies of ovary, breast, colon, lung, pancreas and liver. In each of these cancer types, the mechanisms leading to malignancy-related ascites may be different. Peritoneal carcinomatosis is a major cause of malignancy-related ascites. Other causes include massive liver metastasis causing portal hypertension, chronic hypoalbuminaemia, hepatocellular carcinoma, chylous ascites from lymphoma and Budd-Chiari syndrome due to occlusion of hepatic veins (Runyon BA, 1988).

In patients with cancer, aside from those who develop ascites as a result of portal hypertension, the benefit of intravenous albumin infusion with large volume paracentesis is uncertain, if at all present. Locally, the current clinical practice is for infusion of intravenous albumin during abdominal paracentesis in patients with malignancy-related ascites regardless of cause. The drawbacks of such an approach include exposing patients to risk of anaphylaxis and increased financial costs (50 ml of 20% Albumin costs $42).

Granted that the potential harms of albumin infusion are rare, the burden of proof to show that an intervention works is held by those who introduce it. To date, there have been no studies specifically examining the role of intravenous albumin infusion in this population. In the setting of advanced cancer where life expectancy is limited, the most clinically relevant benefit of albumin infusion would be to reduce the rates of post-paracentesis circulatory dysfunction. Through a pilot study, we hope to evaluate the effectiveness of IV albumin in reducing rates of hypotension, thereby guiding clinical practice in this area.

Rationale and justification for the Study:

Hypothesis: Intravenous albumin infusion during abdominal paracentesis does not prevent hypotension in patients with malignancy-related ascites without portal hypertension.

Rationale for the Study Purpose:

Three significant outcomes have been proven for the use of intravenous albumin in large volume paracentesis in patients with cirrhosis. These are prevention of hypotension, prevention of hyponatraemia and survival benefit. Ascites in the setting of patients with malignancy usually occurs in advanced stage, of which the most meaningful outcome would be that of prevention of hypotension. At present, the current clinical practice locally is extrapolated from studies in patients with cirrhosis, and some physicians would opt to administer IV albumin with every litre of ascitic fluid drained. We propose a study to compare the rates of hypotension in patients who received IV albumin and those who do not. In this study, we will randomise patients with a known history of cancer who are admitted for symptomatic ascites to two groups. Both groups of patients will undergo insertion of abdominal drain for symptomatic relief. Group 1 will receive intravenous albumin and Group 2 will not.

Rationale for Doses Selected:

In Group 1, 50 ml of 20% intravenous albumin will be given for every litre of ascitic fluid drained as this is the current local preparation and practice.

Rationale for Study Population:

Replacement of intravenous albumin has been established in patients with ascites drainage for patients with liver cirrhosis. It has not been shown to benefit patients with malignancy.

Rationale for Study Design:

There have been no previous studies in patients of this population. This is a prospective pilot randomised study in order to compare the rates of hypotension between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years old
* Inpatients admitted to medical oncology service with symptomatic ascites and who are scheduled for abdominal paracentesis
* Known underlying malignancy
* Blood pressure before abdominal paracentesis more than 90/50 mmHg

Exclusion Criteria:

* Patients with known portal hypertension, defined by serum albumin: ascites gradient (SAAG) more than 11.1 mmol/L, based on previous results in last 1 year
* Patients with a known history of hypotension when getting paracentesis
* Pregnant women

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rates of hypotension | For 48 hours since start of drainage

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernardi M, Caraceni P, Navickis RJ, Wilkes MM. Albumin infusion in patients undergoing large-volume paracentesis: a meta-analysis of randomized trials. Hepatology. 2012 Apr;55(4):1172-81. doi: 10.1002/hep.24786. PMID 22095893
- [Background] Grabau CM, Crago SF, Hoff LK, Simon JA, Melton CA, Ott BJ, Kamath PS. Performance standards for therapeutic abdominal paracentesis. Hepatology. 2004 Aug;40(2):484-8. doi: 10.1002/hep.20317. PMID 15368454